CLINICAL TRIAL: NCT06200584
Title: Synergistic Effect of Vitamin E & D in Reducing the Risk of Effects Associated With Atypical Antipsychotics
Brief Title: Synergistic Effect of Vitamin E & D in Reducing Risk of Effects Associated With Atypical Anti-psychotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Rabia Arshad (Other)
Responsible Party: Sponsor-Investigator, Dr Rabia Arshad, Professor, University of Karachi
Organization: University of Karachi (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: UKarachi2
Record Dates: First submitted 2023-11-21; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Antipsychotics and Neuroleptics Toxicity
MeSH Terms: interventions — Risperidone; Antipsychotic Agents; Olanzapine; Quetiapine Fumarate; Vitamin D; Vitamin E; Vitamins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): normal healthy individuals
- psychotic patients (Experimental): treatment given
  Interventions: Drug: Risperidone; Drug: Olanzapine; Drug: Quetiapine; Drug: Risperidone and Vitamin D and Vitamin E; Drug: Olanzapine and Vitamin D and Vitamin E; Drug: Quetiapine and Vitamin D and Vitamin E

INTERVENTIONS:
Drug: Risperidone — Antipsychotic Agent
  Other Names: neuroleptics
  Arms: psychotic patients
Drug: Olanzapine — Antipsychotic Agent
  Other Names: neuroleptics
  Arms: psychotic patients
Drug: Quetiapine — Antipsychotic Agent
  Other Names: neuroleptics
  Arms: psychotic patients
Drug: Risperidone and Vitamin D and Vitamin E — vitamin
  Other Names: vitamin
  Arms: psychotic patients
Drug: Olanzapine and Vitamin D and Vitamin E — vitamin and Antipsychotic agent
  Other Names: vitamin
  Arms: psychotic patients
Drug: Quetiapine and Vitamin D and Vitamin E — Vitamin and Antipsychotic agents
  Other Names: vitamin
  Arms: psychotic patients

SUMMARY:
Atypical antipsychotic drugs are commonly used to treat psychiatric illnesses but they are significantly associated with side effects including acute dystonia, akathisia, parkinsonism (rigidity and tremor), tardive dyskinesia, bradycardia, hypotension, impotence, sleepiness, seizures, severe dreams or nightmares, and hyperprolactinaemia. Vitamin D and E, have been the focus of much research in the past fifteen years, which has revealed multiple roles in the development and function of the body. According to mounting data from the domains of epidemiology and neuroscience, vitamin D and E deficiency have been related to a number of neuropsychiatric issues as well as neurodegenerative diseases. Additionally, antioxidants like vitamin E help to prevent inflammation and highly reactive oxygen molecules from damaging normal cells. The use of vitamin E and D supplements has been suggested to improve the overall outcomes of psychiatric illnesses and neurological diseases. However, the synergistic effect of vitamins E and D in reducing the risk of the adverse effects associated with atypical antipsychotics and improvement in psychiatric illness is not well understood. Therefore, this study was designed to investigate the potential synergistic effect of vitamin E and D supplements for reducing the adverse effects associated with atypical antipsychotics.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Patients using antipsychotic medications such as quetiapine, olanzapine, or risperidone 3. Participants who are between the ages of 20 - 70 years 3. Both gender patients male and female 4. Patients with no other chronic morbidity

ELIGIBILITY:
Inclusion Criteria:

1. Those using antipsychotic medications such as quetiapine, olanzapine, or risperidone.
2. Participants who are between the ages of 20 - 70 years are both sex male and female
3. participants who are taking a combination of one or two antipsychotics.
4. Participants who were under antipsychotic therapy and not diagnosed with type 2 diabetes mellitus.

Exclusion Criteria:

1. Patients at mental hospitals are mostly women who are either pregnant or nursing.
2. Patients who were taking anticonvulsants, ketoconazole, or corticosteroids, or who had a history of other mental or neurologic illnesses, as well as those who used phosphor, calcium, vitamin D supplements or teriparatide, were not included in the study.
3. Participants were also ruled out if they had preexisting conditions including renal or hepatic failure or a parathyroid disease

   -

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Glutathione Peroxidase | 6months
  Serum levels of Glutathione Peroxidase would be determined in each group using a colorimetric approach and commercially available kits because both enzymes are commonly involved in the response to oxidative stress in tissue.(GPX ELISA kit )
Lipid Profile total cholesterol | 6months
  The lipid profile includes the measurement of total cholesterol level in the blood
anti inflammatory markers gamma interferon | 6months
  Expression levels of interferon gamma are determined by polymerase chain reaction. Primers specific to TNF- and IFN- were designed and synthesized for use in polymerase chain reaction (PCR) copy synthesis.
Superoxide Dismutase Activity | 6 months
  Superoxide Dismutase were determined in each group using a colorimetric approach and commercially available kits
lipid profile TG | 6 months
  The lipid profile includes the measurement of triglycerides level in the blood
lipid profile HDL | 6 months
  The lipid profile includes the measurement of high density lipoproteins in the blood
lipid profile VLDL | 6 months
  The lipid profile includes the measurement of very low density lipoprotein levels level in the blood
anti inflammatory markers TNF alpha | 6 months
  Tumor necrosis factor alpha expression is determined by polymerase chain reaction.

SECONDARY OUTCOMES:
Assessment of Psychiatric Improvement, Brief Psychiatric Rating Scale (BPRS) | 6month
  The Brief Mental Rating Scale (BPRS) is a frequently used measure in psychiatry for assessing the severity of various mental symptoms. It is intended to assess the psychological and behavioral features of those suffering from mental health issues. The BPRS is made up of 18 components, each reflecting a different symptom domain. maximum score 168 and minimum score 24

CONTACTS AND LOCATIONS:
Overall Officials: DR MUHAMMAD ABID, MBBS, Principal Investigator — BMSI, JINNAH POST GRADUATE MEDICAL CENTRE,Karachi,Pakistan
Locations (1):
- Jinnah Post Graduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nwosu BU, Meltzer B, Maranda L, Ciccarelli C, Reynolds D, Curtis L, King J, Frazier JA, Lee MM. A potential role for adjunctive vitamin D therapy in the management of weight gain and metabolic side effects of second-generation antipsychotics. J Pediatr Endocrinol Metab. 2011;24(9-10):619-26. doi: 10.1515/jpem.2011.300. PMID 22145446
- [Background] de Bartolomeis A, Ciccarelli M, Vellucci L, Fornaro M, Iasevoli F, Barone A. Update on novel antipsychotics and pharmacological strategies for treatment-resistant schizophrenia. Expert Opin Pharmacother. 2022 Dec;23(18):2035-2052. doi: 10.1080/14656566.2022.2145884. Epub 2022 Nov 17. PMID 36368055
- [Background] Nagashima T, Shirakawa H, Nakagawa T, Kaneko S. Prevention of antipsychotic-induced hyperglycaemia by vitamin D: a data mining prediction followed by experimental exploration of the molecular mechanism. Sci Rep. 2016 May 20;6:26375. doi: 10.1038/srep26375. PMID 27199286
- [Background] Yuan T, Wang S, Le J, Li Y. Effects of Atypical Antipsychotics on Neuroactive Vitamins in Patients With Schizophrenia. J Clin Pharmacol. 2020 Oct;60(10):1355-1361. doi: 10.1002/jcph.1625. Epub 2020 May 19. PMID 32428979

DOCUMENTS (3):
  • Study Protocol: cover letter (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT06200584/Prot_000.pdf
  • Study Protocol: cover letter (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT06200584/Prot_001.pdf
  • Informed Consent Form (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT06200584/ICF_002.pdf